CLINICAL TRIAL: NCT02947425
Title: TARGIT R: TARGeted Intraoperative radioTherapy (TARGIT) Registry Database
Brief Title: TARGeted Intraoperative radioTherapy (TARGIT) Registry Database
Acronym: TARGIT R
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: TARGIT R; ISRCTN91179875 (Other: ISRCTN registry); 14/LO/1452 (Other: UK NRES)
Record Dates: First submitted 2016-08-15; First posted 2016-10-27 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Early-Stage Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospectively registered database of patients with early breast cancer who will be treated with radiotherapy during surgery. More than 2000 women have already received this treatment in clinical trials. This study will monitor the health status of women who receive this treatment outside of a clinical trial, especially those who might not have been eligible for the original clinical trials. The aim is to confirm the long-term effectiveness and safety of the technique.

DETAILED DESCRIPTION:
Registration of patients selected for this treatment; collecting data regarding safety and toxicity on patients who have had treatment with TARGIT.

Outcomes will be measured over short and long terms. Outcome measures will include effectiveness and safety, assessed in various cohorts of patients. Core outcomes will be used for effectiveness. In addition, true recurrence (basically, ipsilateral breast tumor recurrence at the same site as the original primary) will be used as defined by Recht. Safety outcomes will be based on Common Toxicity Criteria.

Budget impact analysis of IORT in subgroups of patients will be assessed. This amounts to using cost data to calculate the mean incremental (or extra) cost per person treated using intraoperative radiotherapy (IORT) versus external beam radiotherapy (EBRT) and mastectomies (where IORT could have been given instead) and then multiplying this by the total patients eligible nationally for IORT, to calculate the total expected budget impact on the NHS if IORT in these subgroups was rolled out nationally.

ELIGIBILITY:
Inclusion Criteria:

* Recommended treatment by MDT
* Consent has been obtained to have patient data to be collected

Exclusion Criteria:

* Pregnancy (females who have a positive pregnancy test prior to surgery)
* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population is very wide, reflecting the pragmatic nature of this study.
  There will be few inclusion and exclusion criteria. Basically, any person aged over 18 with early breast cancer suitable for breast conserving surgery will be eligible. More specific entry criteria for those aged 45 or less will be defined by a participating institution's multidisciplinary team. Experience to date has indicated that there are many patients who are deemed unsuitable for a course of external beam radiotherapy whose only option is therefore mastectomy; such situations can be difficult to define in advance, and should be decided on a case-by-case basis.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2013-07; Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Local tumour control (defined as no recurrent tumour in the ipsilateral breast) | Five years
  Confirmation that the TARGIT technique results in an acceptably low rate of local recurrence when given outside of a randomised controlled trial.
Adverse events related to the primary treatment of the breast cancer. | Five years
  Confirmation that the TARGIT technique results in an acceptably low rate of safety events assessed by CTCAE v4.0 when given outside of a randomised controlled trial.

SECONDARY OUTCOMES:
Cost effectiveness | Five years
  Confirmation that the TARGIT technique is cost-effective as assessed by both health related quality of life (EQ5D) and cost data.

CONTACTS AND LOCATIONS:
Overall Officials: Jayant S Vaidya, Principal Investigator — UCL
Locations (3):
- United Kingdom (3):
  - Royal Free Hospital, London
  - The London Clinic, London
  - Royal Hampshire County Hospital, Winchester

IPD SHARING:
Plan to Share IPD: Yes
All requests for data sharing will adhere to the UCL Surgical & Interventional Trials Unit (SITU) data sharing agreement policy. UCL Medical School is supportive of data sharing and will endeavour to assist in requests for data sharing. These data will be held at UCL on secure servers and will not be released to any third parties until the final study report has been published. All requests for access to the data will be formally requested through the use of a SITU data request form which will state the purpose, analysis and publication plans together with the named collaborators. All requests are dealt with on a case by case basis. All requests will be logged and those successful will have a data transfer agreement which will specify appropriate acknowledgement of the Royal Free Hospital, the sponsor, and funders.